CLINICAL TRIAL: NCT02011477
Title: Comparison of Hypoalgesic Effects of Neural Stretching Versus Neural Gliding: a Randomized Clinical Trial
Brief Title: Hypoalgesic Effects Neural Mobilization Techniques
Acronym: NM
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Josue Fernandez Carnero (Other)
Collaborators: Universidad Autonoma de Madrid (Other)
Responsible Party: Sponsor-Investigator, Josue Fernandez Carnero, Associate Professor, Universidad Rey Juan Carlos
Organization: Universidad Rey Juan Carlos (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSEULS-PI-001/2013
Record Dates: First submitted 2013-12-02; First posted 2013-12-13 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2013-12

CONDITIONS: Hyperalgesia
Keywords: Neural mobilization; Physical therapy; Asymptomatic subjects
MeSH Terms: conditions — Hyperalgesia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Neural glide (Experimental): This technique involves two movements, initial and final. It consists of going from one to the other constantly. The therapist took the subject's head by putting his hands on the suboccipital and front region. In the initial movement, the therapist perform craniocervical flexion in the subject, while he helped with his right elbow to rectify the dorsal spine of the subject; at the same time, the subject perform dorsiflexion of the right ankle. In the final movement, the subject must increase thoracic kyphosis at the same time as perform plantarflexion in the right ankle; also, the therapist performed craniocervical extension in the subject. The session lasted 7 minutes.
  Interventions: Other: Neural stretching
- Placebo (Placebo Comparator): The model of the ultrasound (ENRAF-NONIUS, P.O. Box 12080, 3004 GB Rotterdam, The Netherlands). The subject was placed in a prone position, with arms along the body and the head in the hole of the examining couch. The therapist applied a non-therapeutic dose of ultrasound for 7 minutes with no break all over the cervical area and trapezius, in circles.
  Interventions: Other: Neural Glide; Other: Neural stretching
- Neural Stretching (Active Comparator): In the start position, the subject was supine on a couch, with knees bent with the right leg above the left, and supported with the popliteal zone. Both hands were crossed over the chest. One hand was placed on the occipital, and the other hand was placed over the crossed hands of the subject . In the final position, the therapist made the subject execute a craniocervical flexion while he pushed the subject's hands against the chest, in order to increase thoracic kyphosis. At the same time, the subject had to raise the elevated leg without separating the popliteal zone in the other knee, while maintaining dorsiflexion of the ankle and a maximum knee extension. The session lasted 7 minutes.
  Interventions: Other: Neural Glide

INTERVENTIONS:
Other: Neural Glide — This technique involves two movements, throughout several joints to glide the nerves. The subject sit on a couch with the right lower limb extended and the left lower limb flexed. The therapist will take the subject's head by putting his hands on the suboccipital and front region. In the initial movement, performe craniocervical flexion in the subject, while he helped with his right elbow to rectify the dorsal spine of the subject; at the same time, the subject performed dorsiflexion of the right ankle. In the final movement, the subject must increase thoracic kyphosis at the same time as performing plantarflexion in the right ankle; also, the therapist performed craniocervical extension in the subject
  Arms: Neural Stretching; Placebo
Other: Neural stretching — In the start position, the subject was supine on a couch, with knees bent with the right leg above the left, and supported with the popliteal zone. Both hands were crossed over the chest. The therapist was on the subject´s side, with his knee below the subject's head, bringing stability. One hand was placed on the occipital, and the other hand was placed over the crossed hands of the subject
  Arms: Neural glide; Placebo

SUMMARY:
The purpose of this study was to evaluate the immediate mechanical hypoalgesic effect of neural mobilization in asymptomatic subjects. We also compared neural gliding versus neural stretching to see which produced greater hypoalgesic effects in asymptomatic subjects.

DETAILED DESCRIPTION:
Asymptomatic subjects will be randomly allocated into three groups: the neural glide group; the neural stretch group; and the placebo group. Each subject will receive one treatment session. Outcome measures included bilateral pressure pain threshold measured at the trigeminal, cervical, and tibialis anterior points, which will assess pre-treatment and immediately post-treatment by a blinded assessor. Three-way repeated measures analysis of variance was used to evaluate changes in pressure pain threshold, with group (experimental or control) as the between-subjects variable and time (pre-, post-treatment) or side (dominant, nondominant) as the within-subjects variable.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic subjects who met the inclusion criterion of being between 18 and 30 years old.

Exclusion Criteria:

* rheumatologic diseases or any type of cancer, cervical surgery in the past, whiplash trauma and undergoing any type of treatment like physical therapy, manual therapy, osteopathy, chiropraxis, acupuncture during the last three months. All patients recruited for the study complained of pain localized in the neck and/or head region. Initial screening was accomplished by telephone and eligible persons attended a evaluation appointment.
* development of systemic or degenerative diseases
* subjects with symptoms of depression according Beck's questionnaire
* pain in any area between the lower back and head in the last 9 months
* traumatic event in the past 12 months
* history of neck or face pain in the last 6 months

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2013-03; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Pressure pain threshold assessment | 5 minutes
  The pressure pain threshold (PPT) is defined as the amount of pressure at which the sense of pressure first changes to pain. A digital algometer (FDX 25, Wagner Instruments, CT, USA) consisting of a rubber head (1 cm2) attached to a pressure gauge was used to measure PPTs. Force was measured in kilograms (kg); therefore, thresholds were expressed in kg/cm2. The protocol will use a sequence of three measurements, with an interval of 30 seconds between them. PPT will assess over bilateral masseter points 1 and 2, the temporalis muscles, the suboccipital muscle, the upper trapezius muscle (midway between C7 and the acromion), and the tibialis anterior muscle (upper third of the muscle belly) by an assessor blinded to the subject's condition.

CONTACTS AND LOCATIONS:
Overall Officials: Hector Beltran, MSc, Principal Investigator — Centro de estudios La Salle. Universidad Autonoma de Madrid
Locations (1):
- Centro superior de Estudios Universitarios La Salle, Madrid, Aravaca, Spain